CLINICAL TRIAL: NCT01156948
Title: Comparison of Vaginal Versus Oral Misoprostol for Nulliparous Women Prior to Operative Hysteroscopy
Brief Title: Misoprostol For Nulliparous Women Before Hysteroscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Feng Lin, the 1st Affiliated Hospital of Wenzhou Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WenzhouMC
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2008-05

CONDITIONS: Cervical Ripening
Keywords: misoprostol; nulliparous; hysteroscopy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vaginal misoprostol (Active Comparator): vaginal misoprostol was administered to this group of nulliparous women
  Interventions: Drug: misoprostol
- oral misoprostol (Experimental): oral misoprostol
  Interventions: Drug: oral misoprostol

INTERVENTIONS:
Drug: misoprostol — 400ug vaginally the day before surgery
  Arms: vaginal misoprostol
Drug: oral misoprostol — 400ug misoprostol orally the day before the surgery
  Arms: oral misoprostol

SUMMARY:
To compare the impact of 400-microgram self-administered vaginal versus self-administered oral misoprostol at home on preoperative cervical ripening in nulliparous women prior to outpatient hysteroscopy.

DETAILED DESCRIPTION:
There is no consensus on the effect of misoprostol on cervical ripening for nulliparous women. The aim of the study is to compare the impact of 400-microgram self-administered vaginal versus self-administered oral misoprostol at home on preoperative cervical ripening in nulliparous women prior to outpatient hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women who are referred to outpatient hysteroscopy and who have given informed consent will be eligible for study recruitment.

Exclusion Criteria:

* women with a known allergy to misoprostol.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
cervical width | one day

SECONDARY OUTCOMES:
side effects | one day

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, Principal Investigator — the 1st affiliated hospital of Wenzhou Medical College
Locations (1):
- the 1st Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China